CLINICAL TRIAL: NCT07355322
Title: Comparison of a 3-step Bonding System (TRANSBOND™ XT) Versus a 2-step System (GC ORTHO CONNECT™) on Demineralization Around Maxillary Orthodontic Brackets: a Randomized Split-mouth Clinical Trial.
Brief Title: Comparison of a 3-step Bonding System (Transbond™ XT) and a 2-step System (GC Ortho Connect™) on Demineralization Around Maxillary Orthodontic Brackets
Acronym: ORTHOCOLLAGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RECHMPL24_0271; 2025-A01740-49 (Other: ANSM)
Record Dates: First submitted 2025-12-10; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Tooth Demineralization; White Spot Lesion; Demineralization; Orthodontic Appliance Complication; Dental Braces Complication
Keywords: White spot lesions; Orthodontic bonding; Enamel demineralization; Transbond XT; GC Ortho Connect; Split-mouth trial; Orthodontic Brackets; Fixed Orthodontic Appliances; Adolescents; Oral Hygiene; Dental Plaque; Orthodontic Adhesives; Bracket detachment; Bracket debonding
MeSH Terms: conditions — Tooth Demineralization; Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transbond™ XT (3-step system) (Active Comparator): Conventional 3-step bonding system applied on one hemi-arch: acid etching, primer application, adhesive placement, and light curing. Serves as control.
  Interventions: Device: Transbond™ XT bonding procedure
- GC Ortho Connect™ (2-step system) (Experimental): Simplified 2-step bonding system applied on contralateral hemi-arch: acid etching followed by adhesive with integrated primer and light curing. Evaluates potential reduction in enamel demineralization.
  Interventions: Device: GC Ortho Connect™ bonding procedure

INTERVENTIONS:
Device: Transbond™ XT bonding procedure — Brackets are bonded to one hemi-arch using the 3-step protocol: 1) acid etching, 2) primer application, 3) adhesive placement and light curing.
  Arms: Transbond™ XT (3-step system)
Device: GC Ortho Connect™ bonding procedure — Brackets are bonded to the contralateral hemi-arch using the 2-step protocol: 1) acid etching, 2) adhesive with integrated primer, followed by light curing.
  Arms: GC Ortho Connect™ (2-step system)

SUMMARY:
White spot lesions (WSLs) are one of the most common adverse effects of fixed orthodontic treatments, affecting up to 97% of patients treated with labial appliances. These early enamel demineralizations, caused by microleakage between enamel and adhesive, can appear as early as the fourth week of treatment. They not only pose aesthetic concerns but also increase the risk of bracket failure.

This randomized split-mouth clinical trial compares two bonding systems : the traditional three-step system (Transbond™ XT) and the simplified two-step system (GC Ortho Connect™) to assess their impact on enamel demineralization around orthodontic brackets. The degree of demineralization will be measured using the Enamel Decalcification Index (EDI) based on intraoral photographs and confirmed with a fluorescence camera (C50 Acteon).

The aim of the study is to determine whether the simplified bonding protocol can reduce clinical time and saliva contamination risk without increasing enamel demineralization, thus offering a potentially more efficient and conservative approach for orthodontic bonding procedures.

DETAILED DESCRIPTION:
Introduction:

White spot lesions (WSLs) (localized, non-cavitated enamel demineralizations) represent one of the most frequent side effects of fixed orthodontic treatments. Clinically visible in up to 97% of patients undergoing labial orthodontic therapy, these lesions can emerge as early as the fourth week of treatment. They result from microleakage at the adhesive enamel interface, which facilitates bacterial colonization and acid production. Beyond their aesthetic impact, WSLs can compromise bracket adhesion and increase the risk of failure

Fixed orthodontic appliances modify the oral ecosystem, favoring plaque accumulation and hindering efficient brushing, particularly around complex elements such as ligatures, brackets, and springs. Consequently, WSLs constitute a significant clinical concern for both orthodontists and dental surgeons, as these lesions can persist five years after treatment completion.

Bonding Systems Under Investigation :

The conventional bonding protocol, Transbond™ XT, involves three steps: etching, primer application, and adhesive placement. Conversely, the GC Ortho Connect™ system integrates the primer directly into the adhesive, simplifying the bonding procedure to a single step following orthophosphoric acid etching. This reduced protocol minimizes saliva exposure time and enhances bonding strength.

Furthermore, GC Ortho Connect™ contains functional monomers such as 10-MDP (10-methacryloyloxydecyl dihydrogen phosphate), which chemically interacts with hydroxyapatite, forming a stable bond resistant to moisture. While some studies suggest this system reduces the risk of contamination and shortens chairside time, others report slightly deeper and larger lesions compared to the conventional three-step approach. Evidence remains contradictory, with several in vitro studies showing no significant difference in enamel quality between the two bonding systems.

Research Hypothesis and Objectives :

This clinical trial aims to determine whether a significant difference exists in enamel demineralization between a three-step (Transbond™ XT) and a two-step (GC Ortho Connect™) bonding system.

- Primary Objective: Compare the degree of enamel demineralization around orthodontic brackets at debonding between the two systems using intraoral photographs (Enamel Decalcification Index, EDI) and fluorescence imaging (C50 Acteon camera).

* Secondary Objectives:
* Assess enamel demineralization before bonding, at 6 months, and at 12 months.
* Compare bracket failure rates throughout treatment.
* Evaluate plaque accumulation using the Silness and Löe plaque index.

Methodology :

A monocentric randomized split-mouth trial will be conducted at the Montpellier Dental Care Center. Each patient will serve as their own control:

One hemi-arch (control) bonded with Transbond™ XT (3-step system).

The opposite hemi-arch (experimental) bonded with GC Ortho Connect™ (2-step system).

Randomization will be stratified by gender and brushing hand dominance to reduce confounding factors. Inclusion criteria target minors aged 10-16 years requiring fixed labial metallic appliances.

The split-mouth design minimizes interindividual variability (e.g., enamel quality, saliva composition, hygiene habits) and increases statistical power. Additionally, enamel demineralization assessment will be conducted by a blinded examiner to ensure unbiased evaluation.

Conclusion :

This study proposes an innovative clinical comparison between two orthodontic bonding systems to assess their effects on enamel demineralization. If the simplified GC Ortho Connect™ system demonstrates similar or superior outcomes to the conventional Transbond™ XT, it could represent a time-saving, contamination-resistant, and more conservative alternative for orthodontic bonding procedures ultimately improving patient safety and clinical efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 10 to 16 years included,
* Patient attending their first dentofacial orthopedics consultation at the Montpellier Dental Care Center, in adolescent or young adult dentition (according to Démogé classification),
* Patient requiring the placement of a bimaxillary multi-bracket treatment and opting for a metallic vestibular technique.

Exclusion Criteria:

* Syndromic patient (all syndromes included, e.g., cleft lip) or with a severe long-term condition (ALD),
* Patient previously treated with a multi-bracket orthodontic treatment using a mixed, lingual, or vestibular technique,
* Any medical condition deemed incompatible with bracket placement by the investigator,
* Patient with severe MIH (molar-incisor hypomineralization) and/or severe demineralization on one or more teeth (including severe amelogenesis imperfecta or dentinogenesis imperfecta),
* Patient with restorations such as metal crowns, ceramic crowns, porcelain-fused-to-metal crowns, inlays, onlays, or amalgam on one or more vestibular surfaces,
* Patient with oral hygiene incompatible with orthodontic treatment,
* Agenesis of lateral incisors,
* Subject already participating in another interventional clinical trial that could interfere with this study,
* Uncontrolled psychiatric disorder,
* Lack of written informed consent from a legal representative after a reflection period,
* Lack of cooperation or difficulty in communication/comprehension, or refusal of participation by the minor,
* Subject with a dependency or employment relationship with the sponsor or investigator,
* Subject participating in another research study with an ongoing exclusion period,
* Subject not affiliated with the French social security system or not a beneficiary of such a system,
* Protected populations according to the French Public Health Code:

Pregnant or breastfeeding women Subjects deprived of liberty (by judicial, administrative decision, or involuntary hospitalization) Subjects under guardianship or curatorship

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Mean Enamel Decalcification Index (EDI) after Debonding | Up to 24 months
  Mean Enamel Decalcification Index (EDI) per maxillary hemi-arch after debonding of fixed orthodontic appliances. The assessment will be performed using intraoral photographs, based on the 0-3 scoring system of the Enamel Decalcification Index (EDI) by Banks & Richmond, 1994, evaluating white spot lesions (WSLs) around maxillary metallic orthodontic brackets (AO groove .022 x .028). Results will be confirmed using a fluorescence intraoral camera.

SECONDARY OUTCOMES:
Mean EDI per Hemi-Arch | Preprocedural
  Mean Enamel Decalcification Index (EDI) per maxillary hemi-arch, using intraoral photographs and fluorescence intraoral camera, to the 0-3 scoring system of the Enamel Decalcification Index (EDI) by Banks & Richmond, 1994.
Mean EDI per Hemi-Arch | 6 months
  Mean Enamel Decalcification Index (EDI) per maxillary hemi-arch, using intraoral photographs and fluorescence intraoral camera, to the 0-3 scoring system of the Enamel Decalcification Index (EDI) by Banks & Richmond, 1994.
Mean EDI per Hemi-Arch | 12 months
  Mean Enamel Decalcification Index (EDI) per maxillary hemi-arch, using intraoral photographs and fluorescence intraoral camera, to the 0-3 scoring system of the Enamel Decalcification Index (EDI) by Banks & Richmond, 1994.
EDI per Tooth | Preprocedural
  Enamel Decalcification Index (EDI) measured per tooth, according to the 0-3 EDI scoring system.
EDI per Tooth | 6 months
  Enamel Decalcification Index (EDI) measured per tooth, according to the 0-3 EDI scoring system.
EDI per Tooth | 12 months
  Enamel Decalcification Index (EDI) measured per tooth, according to the 0-3 EDI scoring system.
EDI per Tooth | Up to 24 months
  Enamel Decalcification Index (EDI) measured per tooth, according to the 0-3 EDI scoring system.
Occurrence of bracket Detachment per tooth | 6 months
Occurrence of bracket Detachment per tooth | 12 months
Occurrence of bracket Detachment per tooth | Up to 24 months
Total number of detachments per tooth | 6 months
Total number of detachments per tooth | 12 months
Total number of detachments per tooth | Up to 24 months
Total number of detachments per patient | 6 months
Total number of detachments per patient | 12 months
Total number of detachments per patient | Up to 24 months
Plaque Index | Preprocedural
  Plaque Index scored 0-3 according to Silness & Loe, measured with a probe N°6
Plaque Index | 6 months
  Plaque Index scored 0-3 according to Silness & Loe, measured with a probe N°6
Plaque Index | 12 months
  Plaque Index scored 0-3 according to Silness & Loe, measured with a probe N°6
Plaque Index | Up to 24 months
  Plaque Index scored 0-3 according to Silness & Loe, measured with a probe N°6

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane BARTHELEMI, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital Montpellier, Montpellier, France